CLINICAL TRIAL: NCT02093793
Title: A Randomized Controlled Study to Evaluate the Safety and Effectiveness of the Precision Spinal Cord Stimulator Systems Adapted for High-Rate Spinal Cord Stimulation
Brief Title: Safety and Effectiveness Study of the Precision SCS Systems Adapted for High-Rate Spinal Cord Stimulation
Acronym: ACCELERATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A4007
Record Dates: First submitted 2014-03-19; First posted 2014-03-21 (Estimated); Results first posted 2020-07-08 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Chronic Pain; Back Pain
MeSH Terms: conditions — Chronic Pain; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Rate Spinal Cord Stimulation (Experimental): PRECISION SCS Adapted for High-Rate SCS
  Interventions: Device: PRECISION SCS Adapted for High-Rate SCS
- Commercial Rate Spinal Cord Stimulation (Active Comparator): PRECISION SCS Adapted for High-Rate SCS
  Interventions: Device: PRECISION SCS Adapted for High-Rate SCS

INTERVENTIONS:
Device: PRECISION SCS Adapted for High-Rate SCS — Comparison of spinal cord stimulation parameters
  Other Names: Boston Scientific PRECISION Spinal Cord Stimulator System

SUMMARY:
To evaluate the safety and effectiveness of the Precision Spinal Cord Stimulator Systems Adapted for High-Rate Spinal Cord Stimulation as an aid in the management of chronic intractable pain

DETAILED DESCRIPTION:
To evaluate the safety and effectiveness of high rate spinal cord stimulation (HR-SCS) therapy as an aid in the management of chronic intractable pain of the trunk using the Boston Scientific (BSC) PRECISION Spinal Cord Stimulator Systems Adapted for High-Rate Spinal Cord Stimulation

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with chronic, intractable pain of the trunk (NRS ≥ 5) which has been refractory to conservative therapy for a minimum of 90 days.
* Be an appropriate candidate for the surgical procedures required in this study based on the clinical judgment of the implanting physician
* Be 22 years of age or older at the time of enrollment
* Be willing and capable of giving informed consent
* Be willing and able to comply with study-related requirements, procedures, and visits

Exclusion Criteria:

* Have a medical condition or pain in other area(s), not intended to be treated with SCS, that could interfere with study procedures, accurate pain reporting, and/or confound evaluation of study endpoints, as determined by the Investigator
* Have evidence of an active disruptive psychological or psychiatric disorder or other known condition significant enough to impact perception of pain, compliance of intervention and/or ability to evaluate treatment outcome, as determined by a psychologist
* Have previous spinal cord stimulation trial or is already implanted with an active implantable device(s) (e.g. pacemaker, drug pump, implantable pulse generator)
* Have a current systemic infection, or local infection in close proximity to anticipated surgical field
* Pregnant or plan to get pregnant during the course of the study or not using adequate contraception.
* Be participating in another clinical study that may influence the data collected for the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2014-03-27 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wallace, M.D., Principal Investigator — University of California, San Diego
Locations (20):
- United States (20):
  - Hope Research Institute, Phoenix, Arizona
  - Coastal Pain & Spinal Diagnostics, Carlsbad, California
  - UCSD Medical Center - Jacobs Medical Center, La Jolla, California
  - San Diego Pain Institute, San Diego, California
  - Compass Research, LLC, Orlando, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Willis-Knighton River Cities Clinical Research Center, Shreveport, Louisiana
  - MAPS Applied Research Center, Edina, Minnesota
  - Mayo Clinic Foundation, Rochester, Minnesota
  - Mercy Medical Research Institute, Springfield, Missouri
  - Hope Research Institute, Las Vegas, Nevada
  - Premier Pain Centers, LLC, Shrewsbury, New Jersey
  - The Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Pacific Sports and Spine, LLC, Eugene, Oregon
  - Pain Consultants of Oregon, Eugene, Oregon
  - Oregon Health Sciences University, Portland, Oregon
  - Oregon Neurosurgery, Springfield, Oregon
  - Precision Spine Care, Tyler, Texas
  - Pacific Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After subjects were enrolled, they were evaluated per study eligibility criteria. Only those who met all criteria proceeded to receive implant and randomized in the study (as applicable).
Groups:
- High Rate SCS Followed by Commercial SCS: High Rate SCS Settings followed by Commercial Settings
- Commercial SCS Settings Followed by High Rate SCS: Commercial SCS Settings followed by High Rate SCS programming settings
- High Rate Settings Only: High Rate settings only
Period: Overall Study
Arm/Group | High Rate SCS Followed by Commercial SCS | Commercial SCS Settings Followed by High Rate SCS | High Rate Settings Only
Started | 98 | 90 | 68
Completed | 91 | 80 | 65
Not Completed | 7 | 10 | 3

BASELINE CHARACTERISTICS:
Population: After subjects were enrolled, they were evaluated per study eligibility criteria. Only those who met all criteria proceeded to receive implant and randomized in the study (as applicable).
Groups:
- Total: Total of all reporting groups
Arm/Group | High Rate SCS Followed by Commercial SCS | Commercial SCS Settings Followed by High Rate SCS | High Rate Settings Only | Total
Number analyzed (Participants) | 98 | 90 | 68 | 256
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (11.6) | 53.6 (13.1) | 58.5 (11.4) | 55.6 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 49 | 27 | 135
  Male | 39 | 41 | 41 | 121
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 3
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 3 | 7 | 17
  White | 83 | 76 | 57 | 216
  More than one race | 0 | 2 | 0 | 2
  Unknown or Not Reported | 6 | 6 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Responders as Determined by the Cumulative Distribution Function (CDF) of Response Rates
Description: Cummulative distribution function (CDF) of response rates from 0% - 100% numerical rating score (NRS) to derive the entire range of possible responder definitions. This allows us to determine the range of success for all responder rates without the need to identify a certain cutoff (for example, use a 50% responder rate).
  A comparison between the two CDF's was performed by comparing the area under the curves since area between CDFs is equal to the mean difference in low back pain reduction for CR-SCS and HR-SCS. Hence, it can be used to estimate the true underlying difference in responder rates between CR-SCS and HR-SCS
Time Frame: 3 months post-activation
Population: Subjects with a successful trial (High rate settings only) or simulated trial responders (High rate SCS followed by Commercial SCS or vice versa)
Measure: Number; unit: probability
Groups:
- Commercial SCS: Commercial SCS (as part of crossover)
- High Rate SCS: High Rate SCS (as part of crossover)
Arm/Group | Commercial SCS | High Rate SCS | High Rate Settings Only
Number analyzed (Participants) | 30 | 38 | 65
probability | 0.47 | 0.53 | 0.4

ADVERSE EVENTS:
Time Frame: All adverse events were collected through end of crossover phase (High Rate SCS followed by Commercial SCS or vice versa group) or up to 3 months post activation (HR settings only group) for subjects who started the study (n = 256)
Description: All adverse events were collected through end of crossover phase (High Rate SCS followed by Commercial SCS or vice versa group) or up to 3 months post activation (HR settings only group) for subjects who started the study (n = 256)
Groups:
- High Rate SCS: High Rate SCS Settings
- Commercial SCS: Commercial SCS Settings
Arm/Group | High Rate SCS | Commercial SCS | High Rate Settings Only
All-Cause Mortality (participants affected / at risk) | 1/188 | 0/188 | 0/68
Serious Adverse Events (participants affected / at risk) | 8/188 | 3/188 | 2/68
Other Adverse Events (participants affected / at risk) | 11/188 | 13/188 | 4/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Rate SCS (N=188) | Commercial SCS (N=188) | High Rate Settings Only (N=68)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pnuemonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0)
Cerebral Heamorhhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0)
Chronic Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0)
Sick Sinus Syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroentritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0)
Chronic Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Implant Site Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ischemic Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Rate SCS (N=188) | Commercial SCS (N=188) | High Rate Settings Only (N=68)
Implant Site Pain (General disorders) | 11 (12) | 0 (0) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 13 (13) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/93/NCT02093793/Prot_SAP_000.pdf